CLINICAL TRIAL: NCT03851601
Title: Immuno-regulatory Profiling of T Cells in Patients With Graft Versus Host Disease Treated With Extracorporeal Photopheresis
Brief Title: Immuno-regulatory Profiling of T Cells in GVHD Treated With Extracorporeal Photopheresis
Status: Completed | Type: Observational
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Shatha Farhan, Principal Investigator, Henry Ford Health System
Other Study IDs: 9101
Record Dates: First submitted 2019-02-20; First posted 2019-02-22 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: GVHD
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples from 15 patients who receive ECP as part of the treatment of GVHD at our institution will be collected. Samples will be analyzed using the flow cytometer
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ECP: Blood samples from 15 patients who receive ECP as part of the treatment of GVHD at our institution will be collected. Samples will be analyzed using the flow cytometer
  Interventions: Other: blood samples

INTERVENTIONS:
Other: blood samples — Blood samples from 15 patients who receive ECP as part of the treatment of GVHD at our institution will be collected. Samples will be analyzed using the flow cytometer

SUMMARY:
Extracorporeal Photopheresis (ECP) has been used as one of the treatments for graft versus host disease (GVHD). Responses were observed in skin, liver, GI tract, mouth, eye and lung. ECP does not cause immune suppression and therefore less risk of infection or relapse of malignancy. However, the exact mechanism of action of this expensive procedure is not fully understood and no predictors of response to ECP are known so far. This reflects the need for a better understanding of GVHD and its response to ECP. Blood samples from 15 patients who receive ECP as part of the treatment of GVHD at our institution will be collected. Samples will be analyzed using flow cytometer

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are recipients of allogeneic stem cell grafts.
2. Patients with the diagnosis of GVHD according to established criteria and physician decides to treat using ECP
3. Patient must have 100% chimerism with the donor
4. No recent donor lymphocyte infusion.
5. Patients must be able to sustain a platelet count and a hematocrit > 20,000/mL and > 27% respectively, with or without transfusions.
6. The absolute WBC must be >1500/mL
7. Patient must be willing to comply with all study procedures.

Exclusion criteria:

1. Patients who are unable to tolerate the volume shifts associated with ECP treatment due to the presence of any of the following conditions: uncompensated congestive heart failure, pulmonary edema, severe asthma or chronic obstructive pulmonary disease, hepatorenal syndrome.
2. Active bleeding.
3. International normalized ration (INR) >2.
4. Patients with known hypersensitivity or allergy to psoralen.
5. Patients with known hypersensitivity or allergy to both citrate and heparin.
6. Patients with co-existing photosensitive disease (e.g. porphyria, systemic lupus erythematosus, albinism) or coagulation disorders.
7. Active, uncontrolled infection

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are recipients of allogeneic stem cell grafts with the diagnosis of GVHD according to established criteria and physician decides to treat using ECP
Sampling Method: Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2014-08-26 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
effect of ECP on Tregs/TH17 ratio | 6 months
  investigate the effect of ECP on Tregs/TH17 ratio using flow-cytometry in patients with GVHD who receive treatment with ECP

CONTACTS AND LOCATIONS:
Locations (1):
- Henry Ford Hospital, Detroit, Michigan, United States